CLINICAL TRIAL: NCT00191828
Title: A Prospective/Parallel Study on Induced Weight Gain During Atypical Antipsychotic Treatment and Its Management With Psychoeducational Programme
Brief Title: A Study on Induced Weight Gain During Atypical Antipsychotic Treatment and Its Management With Psychoeducational Programme
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7399; F1D-IT-HGLE
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — Olanzapine

INTERVENTIONS:
Drug: olanzapine

SUMMARY:
Olanzapine is an atypical antipsychotic agent indicated for the treatment of schizophrenia and moderate to severe manic episode.

Olanzapine is among the many antipsychotic agents associated with weight gain . The mechanism for antipsychotic drug-related weight gain is not known, although antagonism of serotonin receptors, especially the 5HT2C , and histamine receptors has been hypothesized.

The purpose of this study is to observe the efficacy of a psychoeducational programme in managing the increased weight as a side effect of the olanzapine treatment.

Interventions to prevent weight gain associated with olanzapine should at least include periodic monitoring and recommendations for changes in diet and physical activity.

This is a phase IV, randomised, parallel study of subjects previously treated with olanzapine as antipsychotic monotherapy, which have shown an increase of B.M.I. >7% from the beginning of antipsychotic treatment (assessed during the routine visits). For the first 12 weeks of the trial approximately 60 outpatients, enrolled in one site during a period of one year, will be randomised in a 1:1 ratio into 2 treatment groups: olanzapine + psychoeducational programme or olanzapine alone. In the following 12 weeks of the study all patients undergo the psychoeducational programme. The efficacy of this programme will be assessed monitoring the mean difference from baseline to endpoint in total body weight and BMI.

ELIGIBILITY:
Inclusion Criteria:

* All patients, previously treated with olanzapine as antipsychotic monotherapy, which have shown a weight gain with an increase of BMI >7% (assessed during the routine visits from the beginning of antipsychotic treatment).
* Male or female subjects at least 18 and no more than 65 years of age.
* Subjects must be considered reliable.
* Each subject must have a level of understanding sufficient to perform all tests and examinations required by the protocol.
* Each patient, (and a patient's legal representative if mandated by local law), must understand the nature of the study and must sign an informed consent document.

Exclusion criteria:

* Serious, unstable illnesses such that death is anticipated within 1 year or intensive care unit hospitalization for the disease is anticipated within 6 months. This includes hepatic (specifically any degree of jaundice), renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic diseases (specifically current agranulocytosis with an absolute neutrophil count <500 mm3).
* Prior treatment with any antipsychotic drugs associated to olanzapine.
* Judged clinically to be at significant suicidal or homicidal risk and/or agitated enough to necessitate use of restraints.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-03; Study Completion 2005-08

PRIMARY OUTCOMES:
To observe the efficacy of a psychoeducational programme in managing the olanzapine-associated weight gain

SECONDARY OUTCOMES:
To study the physical and chemical changes induced by weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speack with your personal physician., Sesto Fiorentino, Florence, Italy